CLINICAL TRIAL: NCT00355797
Title: CLEAR: Cylos Pacemaker Responds With Physiologic Rate Changes During Daily Activities
Brief Title: Effectiveness of Pacemaker With Closed Loop Stimulation Compared to Pacemakers With and Without Standard Rate Response
Acronym: CLEAR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biotronik, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20060536
Record Dates: First submitted 2006-07-21; First posted 2006-07-25 (Estimated); Results first posted 2011-06-27 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: Bradycardia
Keywords: Bradycardia; Sinus Node Dysfunction; Chronotropic incompetence; Pacemaker; Rate adaptive
MeSH Terms: conditions — Bradycardia; Sick Sinus Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Closed Loop Stimulation (CLS) (Active Comparator): Pacemaker programmed with Closed Loop Stimulation rate adaptive technology for long-term follow-up data collection.
  Interventions: Device: Closed Loop Stimulation (CLS)
- Standard Rate Adaptive Technology (R) (Active Comparator): Pacemaker programmed with standard rate adaptive technology (R, accelerometer) for long-term follow-up data collection.
  Interventions: Device: Standard Rate Adaptive (R) Technology
- Non-rate adaptive pacing (DDD) (Active Comparator): Pacemaker programmed with no rate adaption (DDD mode) for long-term follow-up data collection.
  Interventions: Device: Non-rate adaptive (DDD) pacing

INTERVENTIONS:
Device: Closed Loop Stimulation (CLS) — Comparison of different pacing modes available on the Cylos pacemaker device. In this intervention group, subjects were programmed to the Closed Loop Stimulation (DDD-CLS or VVI-CLS) pacing mode for the long-term follow-up portion of this study.
  Other Names: Cylos Pacemaker
  Arms: Closed Loop Stimulation (CLS)
Device: Standard Rate Adaptive (R) Technology — Comparison of different pacing modes available on the Cylos pacemaker device. In this intervention group, subjects were programmed to the standard are adaptive pacing mode (DDDR or VVIR) for the long-term follow-up portion of this study.
  Other Names: Cylos pacemaker
  Arms: Standard Rate Adaptive Technology (R)
Device: Non-rate adaptive (DDD) pacing — Comparison of different pacing modes available on the Cylos pacemaker device. In this intervention group, subjects were programmed to the non-rate adaptive pacing mode (DDD or VVI) for the long-term follow-up portion of this study.
  Other Names: Cylos pacemaker
  Arms: Non-rate adaptive pacing (DDD)

SUMMARY:
This is a randomized, prospective, single-blinded, multi-center study involving approximately 1500 patients at 100 centers. The purpose of this study is to demonstrate the effectiveness of Closed Loop Stimulation (CLS) rate adaption technology over both standard rate responsive technology (R) and non-rate responsive mode (DDD) during activities of daily living (ADL).

DETAILED DESCRIPTION:
All patients enrolled in the CLEAR study are implanted with a Cylos pacemaker with Closed Loop Stimulation (CLS) rate adaption technology. Any legally marketed pacing leads may be implanted with the Cylos family of pacemakers.

Prior to enrollment, patients provide written informed consent and are screened to ensure they are eligible to participate in the study. Patients enrolled in the study must have been implanted within 45 days prior to enrollment or are being considered for implant. Once enrolled and implanted with the Cylos pacemaker, the first 500 patients have 45 days to complete an ADL Testing visit. At the Activities of Daily Living (ADL) testing visit, each of the first 500 enrolled patients performs a 6-minute walk test, orthostatic test, and sweep test in three pacing modes, CLS (DDD-CLS or VVI-CLS), standard rate response (DDDR or VVIR) and non-rate responsive mode (DDD or VVI). The order of the pacing modes for testing is randomized in a 1:1:1 ratio. The study primarily analyzes the number of ADL repetitions performed during the 6-minute walk and sweep tests, pulse pressure during the orthostatic test, and secondarily analyzes heart rates during all three tests to compare CLS to both rate responsive and non-rate responsive pacing modes.

For all enrolled patients, the study collects additional data over a 12-month period. Patients are randomized and their pacemaker programmed to one of three pacing modes, CLS, R, or no-rate response in a 2:1:1 ratio, respectively. The patients are then followed for a period of 12 months after the ADL testing (first 500 enrolled patients) or enrollment (patients 501 through 1500). The study collects the following secondary measures to compare CLS to both rate responsive and non-rate responsive pacing modes: changes in 6-minute walk test distance, quality of life, mode reprogramming, atrial fibrillation (AF) burden, cardiac symptoms, and New York Heart Association (NYHA) classification.

ELIGIBILITY:
Inclusion Criteria:

* Implanted within the last 45 days or being considered for implant with a BIOTRONIK pacemaker utilizing CLS rate adaptation technology (currently the Cylos family of pacemakers).
* Ability to give written informed consent
* Geographically stable and able to return for regular follow-ups for 12 months after ADL testing
* At least 18 years old

Exclusion Criteria:

* Patients physically limited and unable to perform all or parts of the ADL testing
* Currently enrolled in any other clinical study
* Patients with medical reasons that preclude regular participation in the follow-ups

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1491 (Actual)
Dates: Start 2006-05; Primary Completion 2008-02 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Freddy Abi-Samra, MD, Principal Investigator — Ochsner Health System
Locations (99):
- United States (99):
  - Raymond Fernandez, Albertville, Alabama
  - Cardiology Associates-Gadsden, Gadsden, Alabama
  - North Alabama Cardiology Center, Gadsden, Alabama
  - Richard Kim, MD, Jasper, Alabama
  - Arizona Heart Institute, Phoenix, Arizona
  - N.R. Devaraj, M.D., Inc., Anaheim, California
  - Family Doctor Medical Group, Benicia, California
  - Caremore Medical Group, Downey, California
  - Multani Medical Group, Downey, California
  - Solano Cardiology, Fairfield, California
  - Pacific Cardiology Associates, Fremont, California
  - San Joaquin General Hospital, French Camp, California
  - Kenny Charn, MD, Jackson, California
  - Kartik Thaker, MD, Lakewood, California
  - Mission Internal Medical Group, Mission Viejo, California
  - Cardio-Pulmonary Associates, Monterey, California
  - St. Luke Cardiovascular Medical Group, Murrieta, California
  - Sacramento Heart & Vascular, Sacramento, California
  - Emad Khaleeli, MD, Torrance, California
  - Torrance Memorial Medical Center, Torrance, California
  - Cardiology Consultants, Turlock, California
  - Ventura Cardiology, Ventura, California
  - Alireza Jafari, MD, Whittier, California
  - Colorado Cardiovascular Center, Boulder, Colorado
  - Boulder Medical Center, Boulder, Colorado
  - Western Cardiology Associates, Denver, Colorado
  - Aurora Denver Cardiology Associates, Denver, Colorado
  - Western Cardiology Associates, Englewood, Colorado
  - Alfieri Cardiology, Newark, Delaware
  - Southern Heart Group, Jacksonville, Florida
  - Melbourne Internal Medicine Associates, Melbourne, Florida
  - Complete Cardiology Care, New Smyrna Beach, Florida
  - Cardiology Consultants, PA, Pensacola, Florida
  - Space Coast Cardiology Consultants, Port Saint John, Florida
  - Brevard Cardiovascular Research Association, Rockledge, Florida
  - Northside Cardiology, PC, Atlanta, Georgia
  - Doris Tummillo, MD, Augusta, Georgia
  - Collins Cardiology, Douglas, Georgia
  - Douglas Medical Specialists, Douglas, Georgia
  - St. Louis Cardiology Consultants - Alton, Alton, Illinois
  - Naeem Khan, MD, Centralia, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Amr El-Shafei, MD, Mount Vernon, Illinois
  - Bluegrass Cardiology, Louisville, Kentucky
  - Tulane University Medical Center, New Orleans, Louisiana
  - Ochsner Clinic, New Orleans, Louisiana
  - New England Cardiovascular Specialists, Boston, Massachusetts
  - West Michigan Cardiology, Grand Rapids, Michigan
  - Thorasic and Cardiovascular Institute, Lansing, Michigan
  - Minneapolis VA, Minneapolis, Minnesota
  - Pidikiti Cardiology, Corinth, Mississippi
  - Coast Heart Institute, Gulfport, Mississippi
  - Midwest Health Professionals, P.C., Bridgeton, Missouri
  - Cardiac Specialists of St. Lukes, Crystal City, Missouri
  - Chand Medical Office, Farmington, Missouri
  - Manzoor Tariq, MD, Festus, Missouri
  - Liberty Cardiovascular Specialists, Liberty, Missouri
  - Heartland Medical Associates, LLC, Moberly, Missouri
  - Lake Cardiovascular Institute, P.C., Osage Beach, Missouri
  - Zia Ahmad, MD, FACC, St Louis, Missouri
  - Gateway Cardiology, PC, St Louis, Missouri
  - St. Louis Cardiology Center, P.C., St Louis, Missouri
  - St. Louis Cardiovascular Center, St Louis, Missouri
  - Lalit Chouhan, MD, St Louis, Missouri
  - St. Louis Heart and Vascular, P.C., St Louis, Missouri
  - Abbas Shehadeh, MD, FACC, West Orange, New Jersey
  - White Sands Institute for Clinical Research, Las Cruces, New Mexico
  - Ohri Medical Group, P.C., Warsaw, New York
  - Heart Group of the Carolinas, Concord, North Carolina
  - Carolina Heart Care, Elkin, North Carolina
  - Carolina Heart Specialists, Gastonia, North Carolina
  - Piedmont Cardiology, Hickory, North Carolina
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Westside Cardiology Associates, Inc., Fairview Park, Ohio
  - Toledo Clinic Cardiology, Toledo, Ohio
  - Oklahoma Heart Institute, Tulsa, Oklahoma
  - Bryan Lucenta, MD, Tulsa, Oklahoma
  - Lakshmi Mizin, M.D., Carbondale, Pennsylvania
  - Alderfer & Travis Associates, Sellersville, Pennsylvania
  - Carolina Heart and Vascular Center, Aiken, South Carolina
  - Charleston Cardiology, Charleston, South Carolina
  - South Carolina Heart Center, Columbia, South Carolina
  - Pee Dee Cardiology, Florence, South Carolina
  - Carolina Heart Specialists, Lancaster, South Carolina
  - Carolina Cardiology Associates, Rock Hill, South Carolina
  - Heart Rhythm Specialists of East Tennessee, Knoxville, Tennessee
  - Lone Star Arrhythmia and Heart Failure Center, Amarillo, Texas
  - Austin Cardiac Clinic, Austin, Texas
  - Fort Worth Heart, Burleson, Texas
  - Dallas VA Medical Center, Dallas, Texas
  - Cardiology Care Consultants, El Paso, Texas
  - Fort Worth Heart, Fort Worth, Texas
  - Cardiology Associates of West Texas, San Angelo, Texas
  - Cardiac Electrophysiology Consultants of S. Texas, San Antonio, Texas
  - Wasatch Cardiology Consultants, PC, Salt Lake City, Utah
  - Cardiovascular Associates of Virginia, Richmond, Virginia
  - McGuire VA Medical Center, Richmond, Virginia
  - Daniel Gottlieb, Burien, Washington
  - Waukesha Heart Institute, Waukesha, Wisconsin

REFERENCES:
- [Derived] Abi-Samra FM, Singh N, Rosin BL, Dwyer JV, Miller CD; CLEAR Study Investigators. Effect of rate-adaptive pacing on performance and physiological parameters during activities of daily living in the elderly: results from the CLEAR (Cylos Responds with Physiologic Rate Changes during Daily Activities) study. Europace. 2013 Jun;15(6):849-56. doi: 10.1093/europace/eus425. Epub 2013 Feb 17. PMID 23419655

RESULTS

PARTICIPANT FLOW:
Groups:
- CLS Rate Adaptive Pacing: Pacemaker programmed with Closed Loop Stimulation (CLS) rate adaptive technology for long-term study follow-up.
- Standard Rate Adaptive Pacing: Pacemaker programmed with standard rate adaptive technology (R, accelerometer) for long-term study follow-up.
- No Rate Adaptive Pacing: Pacemaker programmed with no rate adaption (DDD) for long-term study follow-up.
Period: Overall Study
Arm/Group | CLS Rate Adaptive Pacing | Standard Rate Adaptive Pacing | No Rate Adaptive Pacing
Started | 741 | 369 | 381
Completed | 501 | 221 | 239
Not Completed | 240 | 148 | 142

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CLS Rate Adaptive Pacing | Standard Rate Adaptive Pacing | No Rate Adaptive Pacing | Total
Number analyzed (Participants) | 741 | 369 | 381 | 1491
Age Continuous [Mean (Standard Deviation); unit: years] | 73.5 (11.7) | 72.5 (12.0) | 72.7 (12.4) | 73.1 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 308 | 178 | 190 | 676
  Male | 433 | 191 | 191 | 815

OUTCOME MEASURES:

1. Primary Outcome: Performance of Activities of Daily Living Tests (6-minute Walk and Sweep)
Description: Six-minute walk test and sweep test results for subjects completing tests in all three pacing modes and requiring at least 80% pacing during both tests in the CLS and R pacing modes. The mean composite of repetitions (six minute walk plus sweep) are presented.
Time Frame: within 45 days of enrollment
Population: Patients requiring at least 80% pacing during both tests in the CLS and accelerometer pacing modes are included.
Measure: Mean (Standard Deviation); unit: repetitions
Arm/Group | CLS Rate Adaptive Pacing | Standard Rate Adaptive Pacing | No Rate Adaptive Pacing
Number analyzed (Participants) | 30 | 30 | 30
repetitions | 19.28 (9.70) | 18.09 (9.36) | 18.05 (9.86)
Statistical Analysis 1: Comparison: CLS Rate Adaptive Pacing vs Standard Rate Adaptive Pacing; The endpoint will compare the composite percent change in ADL performance for patients while their devices are programmed to CLS and accelerometer pacing modes, using the no rate adaptive pacing mode as the baseline. Null hypothesis: mean composite of percent change for patients with their device programmed to CLS is less than or equal to the mean composite of percent change for the same patients with their device in accelerometer; Test type: Superiority or Other; p = 0.004, t-test, 2 sided; Mean Difference (Net) = 9.17, 95% CI 2-sided [3.24 to 15.11], Standard Deviation 15.90

2. Secondary Outcome: Change in Quality of Life
Description: Change in Quality of life (QOL) score was determined from baseline to the 12 month follow-up visit. The QOL utilized the physical functioning scale of the SF-36 v2, in which a higher score indicates a better health perception. Best possible score was 57.03 while the worst possible score was 14.94.
Time Frame: baseline and 12 months
Population: Subjects completing a QOL at both baseline and 12 month follow-up were included in an intention to treat analysis.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | CLS Rate Adaptive Pacing | Standard Rate Adaptive Pacing | No Rate Adaptive Pacing
Number analyzed (Participants) | 464 | 208 | 221
score | -0.41 (10.38) | 0.37 (10.38) | -0.41 (9.35)

3. Secondary Outcome: Mode Reprogramming
Description: Number of subjects with device reprogramming from dual (atrial and ventricular pacing) to single chamber (ventricular pacing only) or from single (ventricular pacing only) to dual chamber (atrial and ventricular pacing) during the 12 month follow-up.
Time Frame: 12 months
Population: Subjects completing at least one follow-up visit were analyzed using intention to treat.
Measure: Number; unit: participants
Arm/Group | CLS Rate Adaptive Pacing | Standard Rate Adaptive Pacing | No Rate Adaptive Pacing
Number analyzed (Participants) | 499 | 221 | 238
participants
  Dual to single chamber | 5 | 2 | 1
  Single to dual chamber | 5 | 0 | 1

4. Secondary Outcome: Atrial Fibrillation (AF) Burden
Description: AF burden was measured at 12 months as the percentage of total atrial beats that are at or above 160 bpm.
Time Frame: 12 months
Population: Percentage of atrial burden was collected for subjects utilizing dual chamber pacing that completing a 12-month follow-up visit.
Measure: Mean (Standard Deviation); unit: percentage of atrial beats
Arm/Group | CLS Rate Adaptive Pacing | Standard Rate Adaptive Pacing | No Rate Adaptive Pacing
Number analyzed (Participants) | 409 | 183 | 212
percentage of atrial beats | 7.54 (20.75) | 5.57 (16.81) | 6.65 (19.86)

5. Secondary Outcome: Cardiac Symptoms
Description: Number of subjects exhibiting each cardiac symptom was determined at the 12 month follow-up visit.
Time Frame: 12 months
Population: All subjects answering questions about current cardiac symptoms at the 12-month visit were included in this intention to treat analysis.
Measure: Number; unit: participants
Arm/Group | CLS Rate Adaptive Pacing | Standard Rate Adaptive Pacing | No Rate Adaptive Pacing
Number analyzed (Participants) | 471 | 209 | 230
participants
  Fatigue | 120 | 51 | 54
  Dizzy Spells | 62 | 31 | 29
  Chest Pains | 32 | 21 | 19
  Weakness | 77 | 30 | 30
  Palpitations | 55 | 30 | 24
  Hypotension | 14 | 7 | 9
  Syncope | 5 | 6 | 5
  Shortness of Breath | 94 | 46 | 47

6. Secondary Outcome: Change in New York Heart Association (NYHA) Class
Description: Number of subjects with improved, no change, or worsened NYHA classification at the 12-month visit, as compared to baseline. NYHA classifications (I to IV) are used to assess the various stages of heart failure, with Class I relating to mild heart failure and Class IV relating to severe heart failure.
Time Frame: baseline and 12 months
Population: Subjects with NYHA classifications at both enrollment and at the 12-month visit were analyzed using intention to treat.
Measure: Number; unit: participants
Arm/Group | CLS Rate Adaptive Pacing | Standard Rate Adaptive Pacing | No Rate Adaptive Pacing
Number analyzed (Participants) | 470 | 201 | 223
participants
  Improved 2 classes | 7 | 0 | 1
  Improved 1 class | 56 | 25 | 16
  No change | 341 | 143 | 166
  Worsened 1 class | 65 | 32 | 40
  Worsened 2 classes | 1 | 1 | 0

7. Secondary Outcome: Change in 6-minute Walk Test Distance
Description: Change in number of 10 foot repetitions between baseline and 12-month visit were examined.
Time Frame: baseline and 12 months
Population: Subjects completing the 6 minute walk at both enrollment and at the 12-month visit were included in intention to treat analysis.
Measure: Mean (Standard Deviation); unit: repetitions
Arm/Group | CLS Rate Adaptive Pacing | Standard Rate Adaptive Pacing | No Rate Adaptive Pacing
Number analyzed (Participants) | 436 | 197 | 203
repetitions | 0.03 (3.63) | 0.41 (3.36) | 0.27 (3.95)

8. Primary Outcome: Pulse Pressure During Activities of Daily Living Tests (Orthostatic Test)
Description: Patients completing the orthostatic test in all three pacing modes and that had at least 80% pacing during the test in the CLS and R pacing modes are included in the analysis. The mean pulse pressure is provided.
Time Frame: within 45 days of enrollment
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | CLS Rate Adaptive Pacing | Standard Rate Adaptive Pacing | No Rate Adaptive Pacing
Number analyzed (Participants) | 56 | 56 | 56
mmHg | 48.13 (12.35) | 50.00 (14.4) | 50.54 (15.23)
Statistical Analysis 1: Comparison: CLS Rate Adaptive Pacing vs Standard Rate Adaptive Pacing; The purpose of endpoint was to evaluate the percent change in pulse pressure during test. The null hypothesis was the mean percent change for patients with their device programmed to CLS is greater or equal to the mean percent change for the same patients with their device in accelerometer; Test type: Superiority or Other; p = 0.552, t-test, 2 sided; Median Difference (Final Values) = -1.42, 95% CI 2-sided [-6.17 to 3.33], Standard Deviation 17.74
Statistical Analysis 2: Comparison: CLS Rate Adaptive Pacing vs No Rate Adaptive Pacing; The purpose of endpoint was to evaluate the percent change in pulse pressure during test. The null hypothesis was the mean percent change for patients with their device programmed to CLS is greater or equal to the mean percent change for the same patients with their device without rate adaptative pacing; Test type: Superiority or Other; p = 0.505, t-test, 2 sided; Median Difference (Final Values) = 1.91, 95% CI 2-sided [-3.80 to 7.63], Standard Deviation 21.34

ADVERSE EVENTS:
Arm/Group | CLS Rate Adaptive Pacing | Standard Rate Adaptive Pacing | No Rate Adaptive Pacing
Serious Adverse Events (participants affected / at risk) | 0/741 | 0/369 | 0/381
Other Adverse Events (participants affected / at risk) | 44/741 | 23/369 | 19/381
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CLS Rate Adaptive Pacing (N=741) | Standard Rate Adaptive Pacing (N=369) | No Rate Adaptive Pacing (N=381)
Cardiac symptoms with Catheterization (Cardiac disorders) | 18 (18) | 8 (8) | 5 (5)
Lead revision (Cardiac disorders) | 6 (7) | 4 (4) | 3 (3)
Non-cardiac procedure performed (Surgical and medical procedures) | 8 (8) | 3 (3) | 5 (5)
Device explants (for any reason) (Cardiac disorders) | 4 (4) | 4 (4) | 2 (2)
Symptomatic arrhythmia requiring ablation (Cardiac disorders) | 3 (3) | 2 (2) | 1 (1)
Change in status requiring device upgrade (Cardiac disorders) | 9 (9) | 2 (2) | 3 (3)
Mitral valve replacement (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Pacemaker pocket revision (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Pacemaker change-out (not device related) (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Other cardiac procedure not captured in other groups (Cardiac disorders) | 4 (4) | 6 (6) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less